CLINICAL TRIAL: NCT03895333
Title: Audiological Profiling in Postmenopausal Women With Osteoporosis
Brief Title: Hearing Loss and Osteoporosis
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, Principal investigator, M.D, Department of Obstetrics and GynecologyR, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2019.01.01
Record Dates: First submitted 2019-03-26; First posted 2019-03-29 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Hearing Loss; Osteoporosis, Postmenopausal
Keywords: Bone mineral density; Postmenopause
MeSH Terms: conditions — Hearing Loss; Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: women with hearing loss and osteoporosis will develop the study group.
  Interventions: Other: Audiological profiling and bone mineral densitometry measurement
- control group: women who have hearing loss but have no osteoporosis will constitute the control group.
  Interventions: Other: Audiological profiling and bone mineral densitometry measurement

INTERVENTIONS:
Other: Audiological profiling and bone mineral densitometry measurement — bone mineral densitometry measurements and hearing test patients, osteoporosis according to whether the hearing test will be analyzed.

SUMMARY:
To compare the audiological profiles in postmenopausal women with and without osteoporosis and to examine the pattern of hearing loss in osteoporotic patients. postmenopausal women will be separated as normal, osteopenic and osteoporotic according to bone mineral densitometry results. The evaluation of hearing test will be done in these groups and the results will be compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Between 45-60 years
* postmenopausal women

Exclusion Criteria:

* Women over 60 years old,
* acute or chronic otitis media,
* ear surgery,
* use of ototoxic drugs,
* congenital hearing loss,
* previous long-term steroid use,
* malignant or benign neoplasm of the brain,
* Patients with a history of exposure to noise were excluded from the study.

Ages: 45 Years to 60 Years | Sex: Female
Age Groups: Adult
Study Population: Postmenopausal women who had hearing test between the ages of 45-60 formed the study group
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-01 (Actual)

PRIMARY OUTCOMES:
hearing test results | 1 week
  hearing test results will be examined; Hearing loss result: test passed or test will be recorded as not passed.
bone mineral densitometry measurements | 1 week
  bone mineral densitometry measurements of patients with hearing test. those with bone loss will be evaluated as osteoporosis.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)